CLINICAL TRIAL: NCT03110289
Title: Fecal Microbiota Transplantation in Patients With Active Ulcerative Colitis: Restoration of the Microbiome Through Superdonor Selection
Brief Title: Restoration of the Microbiome Through Superdonor Selection
Acronym: RESTORE-UC
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Fund for Scientific Research, Flanders, Belgium (Other)
Responsible Party: Principal Investigator, Clara Caenepeel, PhD-student under supervision of Prof. Dr. Séverine Vermeire, Universitaire Ziekenhuizen KU Leuven
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: S59525
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Last update posted 2018-03-30 (Actual); Status verified 2018-03

CONDITIONS: Ulcerative Colitis
Keywords: Fecal microbiota transplantation
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Intervention Model Description: We will randomly allocate 108 patients with active ulcerative colitis (Mayo score 4-10, endoscopic Mayo score 2 or 3) in a 1:1 ratio, using a pre-established randomization list, to either 'superdonor' faecal microbiota transplantation or autologous fecal microbiota transplantation (=sham)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Superdonor FMT (Experimental): Fecal microbiota transplantation from a healthy donor that was selected based on a fecal/blood screening, medical interview and on abundance of taxa of the investigators their interest
  Interventions: Other: superdonor FMT
- Autologous FMT (Sham Comparator): Fecal microbiota transplantation derived from feces from the patient her/himself.
  Interventions: Other: autologous FMT

INTERVENTIONS:
Other: superdonor FMT — Fecal microbiota transplantation (FMT) is the transfer of feces from a healthy "superdonor" to the patient.
  Arms: Superdonor FMT
Other: autologous FMT — Fecal microbiota transplantation (FMT) with feces from the patient him/herself
  Arms: Autologous FMT

SUMMARY:
The AIM of this study is to investigate whether the FMT success rate in active UC patients can be increased by intensive donor pre-screening, anaerobic preparation of the FMT and by repeated FMT.

The investigators will start a national multi-centre double-blind randomized sham-controlled trial in April 2017 at 6 hospitals in Belgium and 2 in The Netherlands. They will randomly allocate 108 patients with active ulcerative colitis (Mayo score 4-10, endoscopic Mayo score 2 or 3) in a 1:1 ratio, using a pre-established randomization list, to either 'superdonor' faecal microbiota transplantation or autologous fecal microbiota transplantation (=sham). Each patient will receive 4 FMT's. At baseline FMT will be performed during sigmoidoscopy. At week 1, 2 and 3, the FMT will be administered through rectal instillation. Each FMT will be derived from one donor. Donors will be pre-selected based on a species richness and abundance of taxa of interest. The primary outcome will be steroid-free clinical and endoscopic remission at week 8 (Mayo score ≤2, all subscores ≤ 1, and ≥1 point reduction in endoscopy subscore). Fecal, blood and mucosal samples and questionnaires will be collected at different time points. 16S rRNA stool analysis will be performed to assess the microbial changes after FMT.

DETAILED DESCRIPTION:
Ulcerative colitis (UC) is a chronic relapsing inflammatory bowel disease (IBD) characterized by a diffuse mucosal inflammation, extending proximally from the rectum and causing symptoms of bloody diarrhea. The complex pathogenesis of IBD remains largely unknown.

Manipulation of the enteric microbiota to restore normobiosis has therapeutic potential in IBD. Fecal microbiota transplantation (FMT), whereby fecal microbiota from a healthy donor is transplanted to a patient, is being studied as therapy for active UC patients. Currently three randomized controlled FMT trials have been published in patients with active ulcerative colitis with increasing success9-11. The investigators feel that the FMT success rate in active UC patients can be improved by solving the remaining pressing questions including the use of selected donors, preparation of the FMT, mode and frequency of administration. The investigators therefore designed a new multicenter interventional study with FMT to specifically answer these questions.

The overall main aims of this project are:

Objective 1: They want to examine whether the FMT success rate in active UC patients can be increased by strictly pre-selecting the donors, by standardizing and optimizing the FMT preparation and by repeated FMT administration.

Objective 2: The investigators want to investigate the temporal and functional changes of the intestinal microbiota of UC patients after FMT

Objective 3: They will try to define host-related predictors for (non-)response to FMT with integration of the genetic susceptibility of the patients and their baseline mucosal gene expression

Study design:

This will be a national multicenter (6 university centers) double blind placebo-controlled randomized clinical trial to evaluate the efficacy and safety of FMT in active UC patients (Mayo endoscopic sub score: 2 or 3 and Total Mayo score: 4-10).

The primary endpoint will be steroid-free clinical and endoscopic remission at week 8 (defined as a total Mayo score of 2 or less, with all Mayo subscores of 1 or less, and at least a 1 point reduction from baseline in the endoscopy subscore).

The secondary endpoints will be the investigation of changes in blood and fecal inflammatory markers before and after FMT (e.g. calprotectin and C-reactive protein (CRP)), steroid-free clinical remission, steroid-free clinical response, steroid-free endoscopic remission and steroid-free endoscopic response.

Assuming a success rate of 40% to achieve mucosal healing at week 8 in the donor FMT arm, a treatment difference of 25% in the autologous FMT arm, a sample size of 49 patients per group is required to obtain a power of 80% and a statistical significance at the 5% level. In addition, considering 10% dropouts, a total of 108 patients will be included. Two interim analysis will be performed after inclusion of respectively 33% and 66% of the sample size (N=108) at week 8.

A data and safety monitoring board (DSMB) can than give advice on adjustment of the sample size or early termination.

Fecal, blood, mucosal samples and questionnaires will be collected by the investigators at different time points.

Baseline fecal samples from donors and baseline mucosal samples together with fecal samples (at start of the study and at weeks 0, 1, 2, 3, 4, 8, 12, 24, 52) from patients will be studied by 16S rDNA sequencing based analysis of microbiota.

The goal of the investigators is to improve FMT success rates by microbial prescreening of the donor and by repeated FMT (4 FMT's/patient).

Prior to FMT, donor stool and blood will be screened for pathogens according to the international consensus guidelines. Furthermore, the investigators will pre-select their donors based on species richness and abundance of taxa of interest.

One donor per ten patients will be used and fecal material will be frozen at -80° until use. Therefore the investigators need at least 15 donors to provide fecal samples during the whole trial, inclusive the open-label faze ( +/- 600 donor samples in total).

To optimize the FMT preparation the investigators will prepare the FMT samples under strict anaerobic circumstances.

To standardize the FMT preparation an absolute cell count of the fecal suspension will be determined after a first dilution.

Repeated FMT will be performed for four times with an interval of 1 week until week 4. At baseline, patients will drink 2L Moviprep (standard preparation), afterwards a sigmoidoscopy will be performed whereby the donor feces solution will be administered through a rectal tube.

At week 1, 2 and 3, the donor feces solution will be administered through rectal instillation without prior water enema.

Open label FMT will be available for all patients in the sham-FMT arm from week 8.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients with currently mild-moderate active ulcerative colitis (defined by endoscopic Mayo sub score 2-3 and a Total Mayo score between 4-10)
* Provide written informed consent to participate as shown by a signature on the consent form.
* Patients on concomitant UC-therapy are allowed if the concomitant treatment is restricted to current treatment and at a stable dose (not in the induction faze).

  * Topical therapy and trial medication is not allowed.
  * A maximum dose of 15mg methylprednisolone.
* Negative coproculture (Salmonella, Shigella, Yersinia, Campylobacter, Entamoeba histoliytica, Clostridium difficile toxins and enteropathogenic E. coli)
* Women need to use reliable contraceptives during participation in the study

Exclusion Criteria:

* Consent not obtained or unable to give informed consent
* Condition leading to profound immunosuppression

  * For example: HIV, infectious diseases leading to immunosuppression, bone marrow malignancies, liver cirrhosis
  * Use of systemic chemotherapy
* Use of antibiotics in the previous 4 weeks
* Surgery: Total colectomy, presence of a stoma or ileo-anal pouch
* Presence of an intra-abdominal fistula
* Colon carcinoma
* Diverticulitis
* Patients who are steroid dependent and requiring >15mg methyl prednisone 2 week before START.
* Detection of a gastrointestinal pathogen on stool analysis
* A diagnosis of Crohn's disease of indeterminate colitis
* Females who are pregnant or actively trying to fall pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-04-30 (Estimated); Study Completion 2019-04-30 (Estimated)

PRIMARY OUTCOMES:
steroid-free clinical remission | Week 8
  defined as a total Mayo score of 2 or less and with all Mayo subscores of 1 or less.
steroid-free endoscopic remission or response | Week 8
  defined as at least a 1 point reduction from baseline in the endoscopy subscore.

SECONDARY OUTCOMES:
the investigation of changes in blood and fecal inflammatory markers before and after FMT | Week 8
  changes in calprotectin and C-reactive protein (CRP)
Steroid-free clinical remission | Week 8
  combined Mayo subscores of 1 or less for rectal bleeding plus stool frequency
Steroid-free clinical response | Week 8
  a decrease of 3 points or more on the Mayo score, a 50% or greater reduction from baseline in combined rectal bleeding plus stool frequency Mayo subscores, or both.
Steroid-free endoscopic response | Week 8
  Mayo endoscopic subscore of 1 or less, with a reduction of at least 1 point from baseline
Steroid-free endoscopic remission | Week 8
  Mayo endoscopy subscore of 0 or 1.

CONTACTS AND LOCATIONS:
Overall Officials: Séverine Vermeire, MD and PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caenepeel C, Deleu S, Vazquez Castellanos JF, Arnauts K, Braekeleire S, Machiels K, Baert F, Mana F, Pouillon L, Hindryckx P, Lobaton T, Louis E, Franchimont D, Verstockt B, Ferrante M, Sabino J, Vieira-Silva S, Falony G, Raes J, Vermeire S. Rigorous Donor Selection for Fecal Microbiota Transplantation in Active Ulcerative Colitis: Key Lessons From a Randomized Controlled Trial Halted for Futility. Clin Gastroenterol Hepatol. 2025 Mar;23(4):621-631.e7. doi: 10.1016/j.cgh.2024.05.017. Epub 2024 May 23. PMID 38788915